CLINICAL TRIAL: NCT05060549
Title: Dopamine D3 Receptor Occupancy in Bipolar Depression by Cariprazine (Vraylar): Evaluating Its Antidepressant Benefit
Brief Title: Dopamine D3 Receptor Occupancy in Bipolar Depression
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Martin Lan, Assistant Professor of Psychiatry at CUIMC, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 8079
Record Dates: First submitted 2021-09-22; First posted 2021-09-29 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — cariprazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cariprazine 1.5 mg (Experimental): Participants will receive 1.5 mg daily of cariprazine (Vraylar) for six weeks
  Interventions: Drug: Cariprazine
- Cariprazine 3 mg (Experimental): Participants will receive 3 mg daily of cariprazine (Vraylar) for six weeks
  Interventions: Drug: Cariprazine

INTERVENTIONS:
Drug: Cariprazine — Participants will receive 6 weeks of cariprazine treatment
  Other Names: Vraylar

SUMMARY:
Bipolar disorder is a common condition that can cause significant disability and risk for suicide. Second generation antipsychotic medications can be used to treat depression in bipolar disorder, yet we do not know how they work. Here, we will use a recently approved medication, cariprazine (Vraylar), to treat participants with bipolar depression. They will have brain imaging with PET scans before and during treatment to understand how the medication may be working. Particularly, we will look at the role of the D3 dopamine receptor.

DETAILED DESCRIPTION:
Bipolar disorder is a common and disabling condition with a high rate of suicide. The depressed phase of the disorder accounts for most of the morbidity and mortality. Only four medications are FDA approved to treat bipolar depression. They all include a second generation antipsychotic (SGA), yet the antidepressant mechanism of SGA's is unknown. Not all bipolar patients respond to these treatments, and they can have problematic side effects. There is therefore a great need to understand these medications' antidepressant mechanism of action in order to design more effective treatment options.

This will be an exploratory occupancy study with cariprazine (Vraylar) in unmedicated participants with bipolar depression (n=8). Participants will have [11C]-(+)-PHNO scans before treatment starts, after three weeks of cariprazine, and after six weeks. Participants will be randomized to two dose groups, 1.5 mg daily (n=4) and 3 mg daily (n=4). These are typical doses of the medication for bipolar depression. Serum levels of cariprazine will be measured at each PET scan.

ELIGIBILITY:
Inclusion Criteria:

1. Capacity to provide consent, and informed consent provided
2. Diagnosis of bipolar I disorder and currently meet criteria for DSM5 major depressive episode
3. Depression at enrollment of sufficient severity to score at least 16 on the first 17 items of the Hamilton Depression Rating Scale when including the atypical depression items addendum
4. Age 18-60 years old
5. Patients who are on antidepressant (SSRI, SNRI or bupropion) or antipsychotic medications at presentation will be included if they have failed that regimen, as defined as not achieving at least partial remission after an adequate dose of medications for at least four weeks. Fluoxetine will not be allowed due to its long half-life. Patients will be able to continue to take other mood stabilizer medications (lamotrigine, lithium, valproate, carbamazepine or oxcarbazepine) if they had not made changes to the dose of those medications within eight weeks of signing consent. Benzodiazepines and hypnotics are allowed throughout the study. If taking stimulant medications, they must be willing not to take these during the study.
6. Females of child-bearing potential must be willing to use an acceptable method of birth control throughout the study; abstinence if it does not require changes to usual behavior, birth control pill, male condom, IUD, dep- provera, norplant, male sterilization or female sterilization are acceptable.
7. Participant is likely to tolerate medication washout if indicated

Exclusion Criteria:

1. Diagnosis of any other major psychiatric disorders such as schizoaffective disorder, current psychotic depression. Any recent drug or alcohol use disorder; within 3 months before the study unless mild. Participant meets DSM5 criteria for manic episode at the time of screening, or has YMRS > 12.
2. Previous failed trial of cariprazine, defined by at least six weeks of treatment at the dose of 1.5 mg per day or more. Experienced intolerable side effects of cariprazine in the past. Taking any medications that are either contraindicated or that have clinically significant drug-drug interactions (such as strong CYP3A4 inducers) with cariprazine, unless there is a plan to stop these as part of the washout.
3. History of clinical deterioration when any of the medications that the participant is taking at presentation have been discontinued in the past if they will be discontinued as part of the washout.
4. First-degree family history of schizophrenia if the participant is less than 33 years old.
5. Significant active physical illness, including blood dyscrasias, lymphomas, hypersplenism, endocrinopathies, renal failure, chronic obstructive lung disease, autonomic neuropathies, peripheral vascular disease, neuromuscular disorder or tardive dyskinesia. Any medical diagnoses that would be a contraindication to cariprazine treatment, including any movement disorders. Any history of a seizure disorder.
6. Actively suicidal, as defined by expressive ideation with a plan and intent for suicide, or developing suicidal ideation that requires immediate medical or treatment intervention.
7. Active lactation
8. Electroconvulsive therapy within the past 6 months
9. Participants who endorse a history of prior head trauma and score 1.5 standard deviations below the mean of Trailmaking A & B test
10. Metal implants, cardiac pacemaker, metal prostheses, metal orthodontic appliances or shrapnel in the body unless there is confirmation that the substance is MRI compatible
11. Current, past or anticipated exposure to radiation, including:

    A. Having been badged for radiation exposure in the workplace B. Participation in nuclear medicine protocols in the past year. However, participants will be eligible if the injected dose and dosimetry of the radiotracer used are known and the cumulative annual exposure of the previous study and this study is lower than the annual limit for research participants defined by FDA (21 CFR 361.1)
12. History of claustrophobia that would prevent participation in imaging scans.
13. Inadequate understanding of English
14. Weight >350 lbs or inability to fit into the MRI scanner

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2026-01-06 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
MADRS | 6 weeks
  Montgomery Asberg Depression Rating Scale; Minimum value 0, Maximum 60; higher values indicate greater depression severity

CONTACTS AND LOCATIONS:
Overall Officials: Martin Lan, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No